CLINICAL TRIAL: NCT05172024
Title: NIH RECOVER: A Multi-site Observational Study of Post-Acute Sequelae of SARS-CoV-2 Infection in Adults
Brief Title: Understanding the Long-term Impact of COVID-19 in Adults (RECOVER)
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 21-01226
Record Dates: First submitted 2021-12-27; First posted 2021-12-29 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: SARS-CoV2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Nasal swabs in freeze medium, blood, saliva, stool and urine.
  For patients undergoing Tier 3 invasive testing through additional consent, or undergoing additional tests as part of routine clinical care, residual samples collected for clinical purposes will whenever possible be collected and sent to the biospecimen core, including: cerebrospinal fluid (CSF), biopsy specimens, bronchoalveolar lavage (BAL), lymph node aspirants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with SARS-CoV-2 Infection
- Participants without SARS-CoV-2 Infection

SUMMARY:
This is a combined retrospective and prospective, longitudinal, observational meta-cohort of individuals who will enter the cohort with and without SARS-CoV-2 infection and at varying stages before and after infection. Individuals with and without SARS-CoV-2 infection and with or without Post-Acute Sequelae of COVID-19 (PASC) symptoms will be followed to identify risk factors and occurrence of PASC. This study will be conducted in the United States and subjects will be recruited through inpatient, outpatient, and community-based settings. Study data including age, demographics, social determinants of health, medical history, vaccination history, details of acute SARS-CoV-2 infection, overall health and physical function, and PASC symptom screen will be reported by subjects or collected from the electronic health record using a case report form at specified intervals. Biologic specimens will be collected at specified intervals, with some tests performed in local clinical laboratories and others performed by centralized research centers or banked in the Biospecimen Repository. Advanced clinical examinations and radiologic examinations will be performed at local study sites with cross-site standardization.

DETAILED DESCRIPTION:
Ambidirectional longitudinal meta-cohort study (combined retrospective and prospective) with nested case-control studies.

ELIGIBILITY:
Inclusion Criteria:

INFECTED COHORT -- ADULTS WITH SUSPECTED SARS-COV-2 INFECTION --

An adult qualifies as having suspected SARS-CoV-2 infection if meeting criteria a, b or c below:

1. Patients who meet the following clinical criteria plus one of the epidemiological criteria:

   Clinical Criteria: Acute onset of fever and cough OR acute onset of any three of more of the following signs or symptoms: fever, cough, general weakness /fatigue, headache, myalgia, sore throat, coryza, dyspnea, anorexia/nausea/vomiting, diarrhea, altered mental status.

   Epidemiological Criteria:
   1. Residing or working in an area with a high risk of transmission of virus: closed residential settings, humanitarian settings such as camp and camp-like settings for displaced persons; anytime within the 14 days before symptom onset; or
   2. Residing or travel to an area with community transmission anytime within the 14 days before symptom onset; or
   3. Working in any health care setting, including within health facilities or within the community; anytime within the 14 days before symptom onset.
2. A patient with severe acute respiratory illness: (acute respiratory infection with history of fever or measured fever of ≥38C°; and cough; with onset within the last 10 days; and requires hospitalization).
3. An asymptomatic person not meeting epidemiologic criteria with a positive SARS-CoV-2 Antigen-RDT.

ADULTS WITH PROBABLE SARS-COV-2 INFECTION --

An adult qualifies as having probable SARS-CoV-2 infection if meeting any one of a-d below:

1. A patient who meets clinical criteria for suspected SARS-CoV-2 AND is a contact of a probable or confirmed case or linked to a COVID-19 cluster;
2. A suspect case with chest imaging showing findings suggestive of COVID-19 disease;
3. A person with recent onset of anosmia (loss of smell) or ageusia (loss of taste) in the absence of any other identified cause;
4. Death, not otherwise explained, in an adult with respiratory distress preceding death AND was a contact of a probable or confirmed case or linked to a COVID-19 cluster

ADULTS WITH CONFIRMED SARS-COV-2 INFECTION --

An adult qualifies as having confirmed SARS-CoV-2 infection if meeting any one of a-d below:

1. Any person with a positive Nucleic Acid Amplification Test (NAAT);
2. Any person with a positive SARS-CoV-2 Antigen-RDT OR positive SARS-CoV-2 antibody test* AND meeting either the probable case definition or suspect criteria A OR B;
3. An asymptomatic person with a positive SARS-CoV-2 Antigen-RDT who is a contact of a probable or confirmed case
4. Any person with a positive SARS-CoV-2 nucleocapsid protein antibody test OR a positive SARS-CoV-2 spike protein antibody test IF not vaccinated

   * (*)This protocol modifies the WHO criterion b to add detectable SARS-CoV-2 antibody as a qualifying test.

UNINFECTED COHORT -- ADULTS WITH NO SARS-COV-2 INFECTION --

* Does not meet WHO criteria for a suspected, probable, or confirmed case of SARS-CoV-2 infection, AND
* Has a documented negative SARS-CoV-2 PCR test from a respiratory specimen in the past, if being enrolled as a post-acute control (see XII.H), AND
* Has a documented negative SARS-CoV-2 PCR test from a respiratory specimen at the time of enrollment/screening, AND
* Has a negative SARS-CoV-2 nucleocapsid protein antibody and spike protein antibody test (spike only if not vaccinated) at the time of enrollment, AND
* Live in the same communities or recruited from the same sources as those in the SARS-CoV-2 infected cohort, AND
* Note: uninfected individuals may participate independent of their vaccination status

Exclusion Criteria:

* Individuals who have not yet reached the age of majority
* Unable to provide consent
* Individuals in hospice care
* Any serious medical condition which would prevent long-term participation
* Individuals participating in the study NIH RECOVER-Pediatric: Understanding the long-term impact of COVID on children and families
* Incarcerated individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Infected: Individuals at least 18 years of age meet WHO criteria for suspected, probable or confirmed SARS-CoV-2 infection on or after March 1, 2020.
  Uninfected: Individuals at least 18 years of age who have never met any of the WHO criteria for suspected, probable or confirmed SARS-CoV-2 infection.
Sampling Method: Non-Probability Sample
Enrollment: 15172 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Incidence of candidate PASC symptoms over time | Up to 4 Years
Prevalence of candidate PASC symptoms over time | Up to 4 Years

SECONDARY OUTCOMES:
Incidence of organ injury | Up to 4 Years
Incidence of clinical disease | Up to 4 Years

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Katz, MD, MS, Principal Investigator — NYU Langone Health; Leora Horwitz, MD, Principal Investigator — NYU Langone Health; Andrea Troxel, ScD, Principal Investigator — NYU Langone Health
Locations (86):
- United States (85):
  - University of Alabama at Birmingham (Pregnancy Cohort), Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of South Alabama, Mobile, Alabama
  - Banner University Medical Center (BUMC) - Phoenix, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California San Francisco (Pregnancy Cohort), San Francisco, California
  - University of California, San Francisco (UCSF), San Francisco, California
  - Stanford University, Stanford, California
  - Denver Health and Hospital Authority, Denver, Colorado
  - University of Colorado Denver, Denver, Colorado
  - Yale School of Medicine (YSM), New Haven, Connecticut
  - ChristianaCare Health System, Newark, Delaware
  - George Washington University, Washington D.C., District of Columbia
  - Howard University, Washington D.C., District of Columbia
  - Kaiser Permanente Georgia, Atlanta, Georgia
  - Morehouse School of Medicine (MSM), Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - University of Hawai'i - Mānoa's John A. Burns School of Medicine, Honolulu, Hawaii
  - University of Illinois at Chicago, Chicago, Illinois
  - Northwestern University, Evanston, Illinois
  - Northshore University HealthSystem, Glenview, Illinois
  - University of Kansas Medical Center (KUMC), Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Louisiana State University - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Louisiana State University (LSU), New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Health System, New Orleans, Louisiana
  - Tulane University, New Orleans, Louisiana
  - MaineHealth, Portland, Maine
  - Tufts Medical Center, Boston, Massachusetts
  - Mass General Brigham - Harvard University, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Harvard Medical School, Boston, Massachusetts
  - Harvard School Of Public Health, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center (BIDMC), Boston, Massachusetts
  - Boston University, Boston, Massachusetts
  - Cambridge Health Alliance (CHA), Cambridge, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center (UMMC), Jackson, Mississippi
  - University Of Nebraska Medical Center, Omaha, Nebraska
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University (Pregnancy), New York, New York
  - Columbia University, New York, New York
  - NewYork-Presbyterian Hospital, Queens, New York
  - University of North Carolina (UNC) at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - WakeMed Health & Hospitals, Raleigh, North Carolina
  - University of North Dakota, Grand Forks, North Dakota
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - University Hospitals MacDonald's Women's Hospital, Cleveland, Ohio
  - Metrohealth System, Cleveland, Ohio
  - The MetroHealth System (Pregnancy Cohort), Cleveland, Ohio
  - The Ohio State University - Wexner Medical Center, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - University of Oklahoma Health Sciences Center (OUHSC), Oklahoma City, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
  - Women & Infants Hospital, Providence, Rhode Island
  - Prisma Health Upstate, Greenville, South Carolina
  - Sanford Health, Sioux Falls, South Dakota
  - St. David's Health Care, Austin, Texas
  - University of Texas Medical Branch (UTMB) Galveston, Galveston, Texas
  - Memorial Hermann Health System, Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - UTMB Health League City Campus Hospital & Clinics, League City, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - McKay-Dee Hospital, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Bateman Horne Center, Salt Lake City, Utah
  - Intermountain Medical Center (Intermountain Healthcare), Salt Lake City, Utah
  - University of Utah, Salt Lake City, Utah
  - University of Utah Health, Salt Lake City, Utah
  - LDS Hospital - Intermountain Healthcare, Salt Lake City, Utah
  - Providence Regional Medical Center Everett, Everett, Washington
  - University of Washington, Seattle, Washington
  - Institute for Systems Biology (ISB), Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
  - Providence Sacred Heart Medical Center, Spokane, Washington
  - West Virginia University, Morgantown, West Virginia
  - Medical College Of Wisconsin, Milwaukee, Wisconsin
- Hispanic Alliance for Clinical and Translational Research, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 9 months and no end date.
Access Criteria: The investigator who proposed to use the data and investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose will have access to the data upon reasonable request. Requests should be directed to RECOVER_CSC@NYULangone.org. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Kulik GL, Zheng T, Jolley SE, Ashktorab H, Brim H, Feuerriegel EM, Hafner JW, Hess R, Horne BD, Hornig M, Johnson B, Kim C, Laiyemo AO, McComsey GA, Nikolich JZ, Reid K, Scherry J, Sherif ZA, Tran HG, Verduzco-Gutierrez M, West S, Erlandson KM; RECOVER Adult Cohort Consortium. Physical Function Differences by COVID-19 Status: A Cross-sectional Analysis From the RECOVER Adult Cohort. Phys Ther. 2025 Jul 1;105(7):pzaf063. doi: 10.1093/ptj/pzaf063. PMID 40302048
- [Derived] Erlandson KM, Geng LN, Selvaggi CA, Thaweethai T, Chen P, Erdmann NB, Goldman JD, Henrich TJ, Hornig M, Karlson EW, Katz SD, Kim C, Cribbs SK, Laiyemo AO, Letts R, Lin JY, Marathe J, Parthasarathy S, Patterson TF, Taylor BD, Duffy ER, Haack M, Julg B, Maranga G, Hernandez C, Singer NG, Han J, Pemu P, Brim H, Ashktorab H, Charney AW, Wisnivesky J, Lin JJ, Chu HY, Go M, Singh U, Levitan EB, Goepfert PA, Nikolich JZ, Hsu H, Peluso MJ, Kelly JD, Okumura MJ, Flaherman VJ, Quigley JG, Krishnan JA, Scholand MB, Hess R, Metz TD, Costantine MM, Rouse DJ, Taylor BS, Goldberg MP, Marshall GD, Wood J, Warren D, Horwitz L, Foulkes AS, McComsey GA; RECOVER-Adult Cohort. Differentiation of Prior SARS-CoV-2 Infection and Postacute Sequelae by Standard Clinical Laboratory Measurements in the RECOVER Cohort. Ann Intern Med. 2024 Sep;177(9):1209-1221. doi: 10.7326/M24-0737. Epub 2024 Aug 13. PMID 39133923
- [Derived] Metz TD, Reeder HT, Clifton RG, Flaherman V, Aragon LV, Baucom LC, Beamon CJ, Braverman A, Brown J, Cao T, Chang A, Costantine MM, Dionne JA, Gibson KS, Gross RS, Guerreros E, Habli M, Hadlock J, Han J, Hess R, Hillier L, Hoffman MC, Hoffman MK, Hughes BL, Jia X, Kale M, Katz SD, Laleau V, Mallett G, Mehari A, Mendez-Figueroa H, McComsey GA, Monteiro J, Monzon V, Okumura MJ, Pant D, Pacheco LD, Palatnik A, Palomares KTS, Parry S, Pettker CM, Plunkett BA, Poppas A, Ramsey P, Reddy UM, Rouse DJ, Saade GR, Sandoval GJ, Sciurba F, Simhan HN, Skupski DW, Sowles A, Thorp JM Jr, Tita ATN, Wiegand S, Weiner SJ, Yee LM, Horwitz LI, Foulkes AS, Jacoby V; NIH Researching COVID to Enhance Recovery (RECOVER) Consortium*. Post-Acute Sequelae of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) After Infection During Pregnancy. Obstet Gynecol. 2024 Sep 1;144(3):411-420. doi: 10.1097/AOG.0000000000005670. Epub 2024 Jul 11. PMID 38991216
- [Derived] Horwitz LI, Thaweethai T, Brosnahan SB, Cicek MS, Fitzgerald ML, Goldman JD, Hess R, Hodder SL, Jacoby VL, Jordan MR, Krishnan JA, Laiyemo AO, Metz TD, Nichols L, Patzer RE, Sekar A, Singer NG, Stiles LE, Taylor BS, Ahmed S, Algren HA, Anglin K, Aponte-Soto L, Ashktorab H, Bassett IV, Bedi B, Bhadelia N, Bime C, Bind MC, Black LJ, Blomkalns AL, Brim H, Castro M, Chan J, Charney AW, Chen BK, Chen LQ, Chen P, Chestek D, Chibnik LB, Chow DC, Chu HY, Clifton RG, Collins S, Costantine MM, Cribbs SK, Deeks SG, Dickinson JD, Donohue SE, Durstenfeld MS, Emery IF, Erlandson KM, Facelli JC, Farah-Abraham R, Finn AV, Fischer MS, Flaherman VJ, Fleurimont J, Fonseca V, Gallagher EJ, Gander JC, Gennaro ML, Gibson KS, Go M, Goodman SN, Granger JP, Greenway FL, Hafner JW, Han JE, Harkins MS, Hauser KSP, Heath JR, Hernandez CR, Ho O, Hoffman MK, Hoover SE, Horowitz CR, Hsu H, Hsue PY, Hughes BL, Jagannathan P, James JA, John J, Jolley S, Judd SE, Juskowich JJ, Kanjilal DG, Karlson EW, Katz SD, Kelly JD, Kelly SW, Kim AY, Kirwan JP, Knox KS, Kumar A, Lamendola-Essel MF, Lanca M, Lee-Lannotti JK, Lefebvre RC, Levy BD, Lin JY, Logarbo BP Jr, Logue JK, Longo MT, Luciano CA, Lutrick K, Malakooti SK, Mallett G, Maranga G, Marathe JG, Marconi VC, Marshall GD, Martin CF, Martin JN, May HT, McComsey GA, McDonald D, Mendez-Figueroa H, Miele L, Mittleman MA, Mohandas S, Mouchati C, Mullington JM, Nadkarni GN, Nahin ER, Neuman RB, Newman LT, Nguyen A, Nikolich JZ, Ofotokun I, Ogbogu PU, Palatnik A, Palomares KTS, Parimon T, Parry S, Parthasarathy S, Patterson TF, Pearman A, Peluso MJ, Pemu P, Pettker CM, Plunkett BA, Pogreba-Brown K, Poppas A, Porterfield JZ, Quigley JG, Quinn DK, Raissy H, Rebello CJ, Reddy UM, Reece R, Reeder HT, Rischard FP, Rosas JM, Rosen CJ, Rouphael NG, Rouse DJ, Ruff AM, Saint Jean C, Sandoval GJ, Santana JL, Schlater SM, Sciurba FC, Selvaggi C, Seshadri S, Sesso HD, Shah DP, Shemesh E, Sherif ZA, Shinnick DJ, Simhan HN, Singh U, Sowles A, Subbian V, Sun J, Suthar MS, Teunis LJ, Thorp JM Jr, Ticotsky A, Tita ATN, Tragus R, Tuttle KR, Urdaneta AE, Utz PJ, VanWagoner TM, Vasey A, Vernon SD, Vidal C, Walker T, Ward HD, Warren DE, Weeks RM, Weiner SJ, Weyer JC, Wheeler JL, Whiteheart SW, Wiley Z, Williams NJ, Wisnivesky JP, Wood JC, Yee LM, Young NM, Zisis SN, Foulkes AS. Researching COVID to Enhance Recovery (RECOVER) adult study protocol: Rationale, objectives, and design. PLoS One. 2023 Jun 23;18(6):e0286297. doi: 10.1371/journal.pone.0286297. eCollection 2023. PMID 37352211
- [Derived] Metz TD, Clifton RG, Gallagher R, Gross RS, Horwitz LI, Jacoby VL, Martin-Herz SP, Peralta-Carcelen M, Reeder HT, Beamon CJ, Bind MA, Chan J, Chang AA, Chibnik LB, Costantine MM, Fitzgerald ML, Foulkes AS, Gibson KS, Guthe N, Habli M, Hackney DN, Hoffman MK, Hoffman MC, Hughes BL, Katz SD, Laleau V, Mallett G, Mendez-Figueroa H, Monzon V, Palatnik A, Palomares KTS, Parry S, Peralta-Carcelen M, Pettker CM, Plunkett BA, Poppas A, Reddy UM, Rouse DJ, Saade GR, Sandoval GJ, Schlater SM, Sciurba FC, Simhan HN, Skupski DW, Sowles A, Thaweethai T, Thomas GL, Thorp JM Jr, Tita AT, Weiner SJ, Weigand S, Yee LM, Flaherman VJ. Researching COVID to enhance recovery (RECOVER) pregnancy study: Rationale, objectives and design. medRxiv [Preprint]. 2023 Apr 24:2023.04.24.23289025. doi: 10.1101/2023.04.24.23289025. PMID 37162923

DOCUMENTS (1):
  • Informed Consent Form (2023-06-15): https://cdn.clinicaltrials.gov/large-docs/24/NCT05172024/ICF_000.pdf